CLINICAL TRIAL: NCT06713720
Title: Remote Ischemic Conditioning for Non-Proliferative Diabetic Retinopathy (RIC-NPDR)
Brief Title: Remote Ischemic Conditioning for Non-Proliferative Diabetic Retinopathy
Acronym: RIC-NPDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuxiang Zhang, MD (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, Xuxiang Zhang, MD, Director of Ophthalmology, Xuanwu Hospital, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFH2024-2-20113; CFH2024-2-20113 (Other Grant/Funding Number: Capital's Funds for Health Improvement and Research)
Record Dates: First submitted 2024-11-21; First posted 2024-12-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Retinopathy; Non-Proliferative Diabetic Retinopathy; Remote Ischemic Conditioning; Diabetes Mellitus, Type 2; Randomized Controlled Trial
Keywords: Non-Proliferative Diabetic Retinopathy; Diabetic Retinopathy; Retinal Neurovascular Unit; Remote Ischemic Conditioning; Randomized Controlled Trial
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning Group (Experimental): Participants in this group will receive remote ischemic conditioning (RIC) therapy. This involves five cycles of 5-minute inflation at 200 mmHg followed by 5-minute deflation, twice daily, for at least five days per week over a one-year period.
  Interventions: Device: Remote Ischemic Conditioning Device
- Sham Remote Ischemic Conditioning Group (Sham Comparator): Participants in this group will receive sham remote ischemic conditioning therapy. This involves the same device with inflation pressure set at 60 mmHg, following identical timing and frequency as the intervention group.
  Interventions: Device: Sham Remote Ischemic Conditioning Device

INTERVENTIONS:
Device: Remote Ischemic Conditioning Device — Participants in this group will use a remote ischemic conditioning device that applies five cycles of 5-minute inflation at 200 mmHg followed by 5-minute deflation on both arms, twice daily, for at least five days per week over one year. The device is designed to enhance retinal oxygenation and reduce hypoxia-related damage.
  Arms: Remote Ischemic Conditioning Group
Device: Sham Remote Ischemic Conditioning Device — Participants in this group will use the same remote ischemic conditioning device set to an inflation pressure of 60 mmHg to simulate the treatment. This placebo intervention follows the same timing and cycle frequency as the active intervention group.
  Arms: Sham Remote Ischemic Conditioning Group

SUMMARY:
The goal of this clinical trial is to evaluate whether remote ischemic conditioning (RIC) is a safe and effective treatment for non-proliferative diabetic retinopathy (NPDR) in adults aged 40-80 years with type 2 diabetes. The study aims to address the limitations of current treatments for NPDR by using RIC, a technique involving repeated cycles of ischemia and hypoxia stimulation to activate protective mechanisms against retinal damage.

The main questions it aims to answer are:

Does RIC improve the Diabetic Retinopathy Severity Score (DRSS) after one year of treatment? Does RIC reduce the incidence of vision-threatening proliferative diabetic retinopathy (PDR)? What are the changes in retinal neurovascular unit parameters, visual acuity, and retinal oxygen saturation after RIC treatment?

Participants will:

Undergo RIC therapy using a specialized device on both upper limbs (or a placebo intervention for the control group) for 1 year.

Complete 5 cycles of RIC or placebo treatment twice daily, 5 days per week. Receive routine care for diabetic retinopathy as per clinical guidelines.

Key outcome measures:

Primary outcome: Change in DRSS from baseline after one year. Secondary outcomes: Incidence of PDR, changes in visual acuity, retinal neurovascular unit measures, retinal oxygen saturation, and serum biomarkers (e.g., VEGF, CRP, IL-6).

This randomized, double-blind, placebo-controlled trial aims to recruit 68 participants to ensure 60 complete the study, accounting for a 13% dropout rate. The findings are expected to provide insights into RIC as a novel intervention for NPDR, reducing blindness risk and supporting future large-scale trials.

DETAILED DESCRIPTION:
Non-proliferative diabetic retinopathy (NPDR) represents an early yet critical stage of diabetic retinopathy, a leading cause of vision loss globally. Despite advancements in medical treatments such as anti-VEGF therapy and laser photocoagulation, there remains a significant gap in safe and effective interventions to halt or reverse NPDR progression. Current therapies often focus on advanced disease stages, leaving early-stage management a challenge.

Remote ischemic conditioning (RIC) introduces a novel, non-invasive approach to NPDR treatment. Based on the concept of "fighting hypoxia with hypoxia," RIC employs intermittent cycles of ischemia and reperfusion in the limbs to trigger endogenous protective mechanisms against hypoxic damage. Experimental studies have highlighted RIC's potential benefits, including enhanced retinal oxygenation, reduced pathological vascular proliferation, and preservation of retinal ganglion cells.

This study is designed as a randomized, double-blind, placebo-controlled clinical trial to evaluate RIC's safety and efficacy in adults aged 40-80 years with mild to moderate NPDR. The trial features meticulous inclusion and exclusion criteria to ensure the reliability of findings. Participants will undergo either RIC or placebo therapy using a specialized device. The RIC group will receive therapy at 200 mmHg inflation pressure, while the placebo group will undergo sham treatment at 60 mmHg. Both treatments will follow the same cycle and frequency, ensuring blinding is maintained.

The study's outcomes include comprehensive assessments of retinal structure and function, systemic biomarkers, and safety metrics. These encompass changes in Diabetic Retinopathy Severity Score (DRSS), retinal neurovascular parameters, visual acuity, and retinal oxygenation. Serum biomarkers such as VEGF, CRP, and IL-6 will provide insights into systemic inflammatory and vascular changes post-treatment.

The findings from this trial are expected to offer preliminary evidence on RIC as a safe and effective intervention for NPDR. This work aims to lay the groundwork for future large-scale studies and provide clinicians with a potential strategy to reduce the burden of diabetic retinopathy and its associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years.
* Diagnosed with Type 2 diabetes mellitus.
* Diagnosed with mild to moderate non-proliferative diabetic retinopathy (NPDR) with a DR Severity Score (DRSS) grade of 20-47D.
* Capable of performing daily activities independently.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Presence of diabetic macular edema (macular thickness > 250 μm).
* Significant eye diseases affecting evaluation, such as high myopia, severe cataract, corneal leucoma, glaucoma, retinal detachment, retinal vein occlusion, congenital eye diseases, ocular tumors, or severe infection.
* History of ocular laser or intraocular surgery.
* Poor imaging quality due to refractive media opacity.
* Contraindication to fluorescein fundus angiography.
* Unstable blood glucose (HbA1c ≥ 8.0%) despite oral antidiabetic drugs.
* Severe diabetes complications within the past 6 months.
* Severe, sustained hypertension (systolic ≥ 180 mmHg or diastolic ≥ 110 mmHg).
* Body mass index (BMI) ≥ 28 kg/m².
* Hepatic or renal insufficiency: Alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of normal. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m². Urine albumin/creatinine ratio ≥ 30 mg/g.
* Myocardial infarction within the past 6 months.
* Neurological diseases such as Alzheimer's, Parkinson's, cerebrovascular disease, intracranial tumor, cerebrovascular malformation, or aneurysm.
* Contraindications to RIC, including one-sided subclavian artery stenosis, upper limb injuries or vascular diseases, or limb deformities.
* Severe systemic diseases, such as malignant tumors with a life expectancy of less than 24 months.
* Known pregnancy or breastfeeding.
* Participation in other experimental clinical studies.
* Any other conditions deemed unsuitable by the investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetic Retinopathy Severity Score (DRSS) | Baseline and 1 year after intervention
  The primary outcome measure is the change in the Diabetic Retinopathy Severity Score (DRSS) from baseline to 1 year after intervention. The DRSS is a standardized grading system used to assess the severity of diabetic retinopathy, with changes reflecting disease progression or improvement.

SECONDARY OUTCOMES:
Incidence of Proliferative Diabetic Retinopathy (PDR) | 1 year after intervention
  The incidence of participants who progress to proliferative diabetic retinopathy (PDR) within one year after the intervention. PDR progression is identified based on clinical examination and fundus photography.
Change in Retinal Neurovascular Unit Parameters | Baseline and 1 year after intervention
  Changes in parameters of the retinal neurovascular unit, including macular capillary densities (superficial and deep), radial peripapillary capillary density, ganglion cell complex thickness, and retinal nerve fiber layer thickness, assessed through optical coherence tomography angiography (OCTA) from baseline to 1 year.
Change in Retinal Oxygen Saturation | Baseline and 1 year after intervention
  The change in retinal oxygen saturation levels measured using retinal oximetry between baseline and 1 year after intervention. Improvements are expected to reflect reduced retinal hypoxia.
Change in Visual Acuity | Baseline and 1 year after intervention
  The change in best-corrected visual acuity (BCVA) measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart between baseline and 1 year after intervention.
Change in Serum Biomarker Levels | Baseline and 1 year after intervention
  The change in serum levels of vascular endothelial growth factor (VEGF), C-reactive protein (CRP), interleukin-6 (IL-6), and occludin from baseline to 1 year. These biomarkers provide insights into systemic inflammation, vascular health, and blood-retinal barrier function.

OTHER OUTCOMES:
Incidence of Local Complications Related to Intervention | Up to 1 year during intervention
  The incidence of experiencing local complications, including upper limb pain, erythema, edema, skin injury, and ischemia, related to the remote ischemic conditioning device during the one-year intervention period.
Retention Rate of Participants | 1 year after intervention
  The retention rate of participants who complete the one-year intervention without withdrawal. This measures feasibility and adherence to the intervention protocol.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No